CLINICAL TRIAL: NCT06154551
Title: Evaluation of the Levels of Salivary Paxillin Oral Premalignant and Malignant Lesions
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Olfat Shaker (Unknown)
Responsible Party: Principal Investigator, Yasmine Kamal, lecturer of oral medicine, Cairo University
Other Study IDs: 321122
Record Dates: First submitted 2023-11-17; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Comparison of Salivary Paxillin Levels in OPMLs and OSCC to Healthy Subjects
Keywords: oral potentially malignant lesions; oral squamous cell carcinoma; saliva; paxillin
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: fifteen patients with OPMLs (lichen planus, leukoplakia)
  Interventions: Diagnostic Test: Paxillin biomarker
- Group B: fifteen patients with OSCC
  Interventions: Diagnostic Test: Paxillin biomarker
- Group C: fifteen systemically healthy control subjects
  Interventions: Diagnostic Test: Paxillin biomarker

INTERVENTIONS:
Diagnostic Test: Paxillin biomarker — Paxillin used as a salivary biomarker

SUMMARY:
This investigation was carried out to analyze and compare the salivary paxillin levels between oral premalignant and malignant lesions (OPMLs), OSCC and the healthy controls in order to assess its potential role as a biomarker of oral cancer aiming for early diagnosis and better prognosis of OSCC.

Methods: Forty-five patients, ranging in age from thirty to seventy-five, were divided into three groups: fifteen patients with OPMLs (lichen planus, leukoplakia), fifteen patients with OSCC, and fifteen controls who were in general well. Paxillin was identified in saliva samples by using an ELISA kit.

DETAILED DESCRIPTION:
The aim of this study is: comparison of salivary paxillin levels in oral premalignant lesions and OSCC to its levels in healthy subjects.

Subjects and Methods Forty-five participants between the ages of 30 and 70 were accepted for this study. They were registered in the outpatient's clinic of Oral Medicine and Periodontology department in Faculty of Dentistry,Cairo university. Three sets of subjects were assigned: fifteen patients with premalignant lesions, fifteen patients with OSCC, and fifteen systemically healthy control subjects. A complete medical history was obtained for each individual using a modified Cornell Medical Index questionnaire. Upon receiving clarification regarding the scope of the inquiry, each participant completed an informed consent form.

Patients with OSCC were clinically diagnosed, and biopsy specimens from the lesions were taken for histology to confirm the diagnosis.

Collection of saliva samples:

Unstimulated Salivary samples were collected once preoperatively before any intervention All participants were asked to refrain from drinking, eating, or chewing gum for at least 60 minutes before sampling. Samples were collected by asking the patient to swallow first, then lean the head forward for 5 minutes and spit the entire saliva into 50-ml sterile centrifuge tubes. After being assembled, all specimens were immediately stored at -20 ºC until tested.

Quantitation of Human Paxillin salivary level:

Saliva was collected from patients and controls. After centrifugation, the supernatant was separated for detection of Paxillin by using the ELISA technique provided by Cloud Clone Corp, Houston, USA, Catalogue Number: E-01184hu. This kit's microtiter plate has been pre-coated with a paxillin-specific antibody. The relevant microtiter plate wells are then treated with a biotin-conjugated antibody specific to paxillin. Then, Avidin conjugated to Horseradish Peroxidase (HRP) is added and incubated in each microplate well. After adding the TMB substrate solution, only the wells containing paxillin, biotin-conjugated antibody, and enzyme-conjugated Avidin will change colour. The enzyme-substrate reaction is stopped by adding a solution of sulphuric acid, and the colour change is measured spectrophotometrically at 450nm 10nm. The samples' optical density (OD) is then compared to the reference curve to determine their paxillin concentration.

Statistical analysis:

Categorical data were given as frequency and percentage values, and Fisher's exact test was used to assess them. Mean and standard deviation (SD) numbers were used to depict numerical data. The Shapiro-Wilk test was used to determine their normalcy. A one-way ANOVA test followed by Tukey's post hoc test was used to analyse normally distributed data (age and Paxillin (ng/mL) levels). ROC curve analysis was done to determine diagnostic accuracy. A z-test was used to compare ROC curves. The significance level was set at p<0.05 for all tests. R statistical analysis software version 4.3.1 for Windows was used for the statistical analysis [18].

ELIGIBILITY:
Inclusion Criteria:

* patients with leukoplakia patients with atropic lichen planus patients with bullous erosive lichen planus patients with squamous cell carcinoma

Exclusion Criteria:

* patients with papular lichen planus patients with underlying systemic disease leukemic patients smokers hepatic patients

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty-five participants between the ages of 30 and 70 were accepted for this study. They were registered in the outpatient's clinic of Oral Medicine and Periodontology department in Faculty of Dentistry,Cairo university. Three sets of subjects were assigned: fifteen patients with premalignant lesions, fifteen patients with OSCC, and fifteen systemically healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
salivary levels of paxillin | once preoperatively
  to detect the levels of salivary paxillin and compare its levels in the three study groups

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine Ramadan, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hussine AA, Selim K, Shaker O, Kamal Y. Evaluation of the levels of salivary paxillin in oral potentially malignant disorders and malignant lesions. BMC Oral Health. 2024 Jul 24;24(1):834. doi: 10.1186/s12903-024-04569-z. PMID 39048985